CLINICAL TRIAL: NCT04646031
Title: Expanded Access Use of T89 in An Intermediate-size Patients Population for the Treatment of Severe "Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2)" Infection Disease Patients (COVID-19)
Brief Title: Expanded Access to T89 for Treatment Use in Intermediate-size Patients Population With COVID-19
Status: No longer available | Type: Expanded Access
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Collaborators: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: T89-ROUSA-01
Record Dates: First submitted 2020-11-24; First posted 2020-11-27 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: Twenty (20) patients with severe COVID-19 as participants
MeSH Terms: conditions — COVID-19 | interventions — T89 herbal drug

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: T89 capsule — T89 capsule, an medicinal product for oral use under active INDs in the US is a botanical drug containing 75mg active substance of the water extract of Danshen and Sanqi.
  Other Names: Dantonic

SUMMARY:
This expanded access use program will provide a botanical drug of T89 for treatment use in an intermediate-size population infected with SARS-CoV-2 who have severe COVID-19, or who are judged by a healthcare provider to be at high risk of progression to severe or life-threatening condition.

DETAILED DESCRIPTION:
T89 capsule is a botanical drug product for oral use. The drug substance of T89 capsule is the water extract of two widely used herb medicines: Danshen (Radix Saliva Miltiorrhize Bge., RSM) and Sanqi (Radix Notoginseng, RN).

A large number of researches have shown that T89 has the effects of activating blood circulation and removing blood stasis. Clinical trials conducted in China and US also show that T89 can significantly improve blood oxygen saturation at high altitudes and alleviate the symptoms of hypoxia. It has been also reported that T89 is effective in treating myocardial ischemic diseases.

Basic studies show that T89 can improve red blood cell oxygen delivery capacity, reduce reactive oxygen species (ROS) related tissue damage, alleviate tissue and organ injuries caused by ischemia by improving microcirculation, improve energy metabolism and increase adenosine triphosphate (ATP) production in myocardial tissue, inhibit the reduction of hematocrit, albumin leakage, neutrophil CD18 and intercellular cell adhesion molecule-1 (ICAM-1), preventing deterioration of microcirculation caused by ischemia and hypoxia, and inhibit platelet aggregation and adhesion.

The objective of this expanded access program is to provide T89 for treatment use in an intermediate-size population with severe COVID-19, with the dosing regimen of 300mg (four T89 capsules) each time, orally, three time daily for 14 days, followed by a follow-up visit by call on Day 21.

ELIGIBILITY:
Inclusion Criteria:

* Was hospitalized due to COVID-19 confirmed by positive testing of standard reverse transcription-polymerase chain reaction (RT-PCR) assay;
* Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥30 per minute, heart rate ≥125 per minute, oxygen saturation by pulse oximetry (SpO2) ≤86% on room air or PaO2/FiO2 <300 (PaO2=Arterial oxygen pressure, FiO2=Inspired oxygen fraction );
* With at least one of following underlying diseases such as hypertension, diabetes, and cardiovascular disease;
* Oxygen therapy is clinically indicated at the start of screening.
* Abnormal low platelet counts and/or other measurements indicative of systemic thrombosis, such as platelet counts <150,000/µL; 0.6 μg/mL< D-dimer ≤2.0 μg/mL (i.e., 1.2-4×upper limit of normal(ULN); ULN=0.5 μg/mL).

Exclusion Criteria:

* Requiring immediate intensive care unit (ICU) administration and treatment.
* Need for high-flow nasal cannula oxygen delivery, noninvasive ventilation, invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO).
* Progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatment.
* Have known congenital hypercoagulopathy including but not limited to factor V Leiden (FVL) homozygous and heterozygous, protein C or protein S deficiency. And patients who have hypercysteinemia.
* Have congenital bleeding disorder including but not limited to von Willebrand disease, hemophilia A (factor VIII deficiency) hemophilia B (factor IX deficiency).
* With alanine aminotransferase (ALT) ≥5×ULN, or aspartate aminotransferase (AST) ≥5×ULN, or alkaline phosphatase (ALP) ≥5×ULN, or Total Bilirubin (TBILI) ≥2×ULN, or platelet counts <50,000/µL, or neutrophil counts <1,000/µL.
* Has severe preexisting pulmonary disease including but not limited to chronic obstructive pulmonary disease (COPD), pulmonary fibrosis, pneumonectomy etc. Subjects with extrinsic restrictive lung disease due to obesity can be enrolled.
* With stage 4 severe kidney failure (i.e. estimated glomerular filtration rate (eGFR) <30) or requiring dialysis.
* With congestive heart failure with New York Heart Association (NYHA).

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Meehan, PhD, MD, Principal Investigator — MultiCare Health System
Locations (1):
- MultiCare Health System, Tacoma, Washington, United States